CLINICAL TRIAL: NCT03628313
Title: Valvular Aortic Stenosis Prognosis Study: Prospective and Retrospective Follow-up of a Cohort of Patients With Aortic Valve Narrowing
Brief Title: Valvular Aortic Stenosis Prognosis Study
Acronym: EPRAoV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2014-16
Record Dates: First submitted 2018-07-31; First posted 2018-08-14 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Morality
Keywords: Echoacrdiography; EchoDoppler; Aortic valve stenosis; Prognosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aortic valve stenosis: The participants will be identified from the Transthoracic ultrasound echocardiography reports of the echocardiography laboratory of the University Hospital of Amiens and CH Philibert for the retrospective part. They are analyzed during echocardiography at the echocardiography laboratory of two participating centers when a diagnosis of aortic stenosis is made. Patients are informed by newsletter.
  Interventions: Other: Transthoracic ultrasound

INTERVENTIONS:
Other: Transthoracic ultrasound — Patients are prospectively identified during echocardiography performed in the echocardiography laboratory of the two participating centers when a diagnosis of aortic stenosis is made.

SUMMARY:
Aortic stenosis is the most common valvulopathy in Western countries. Cardiac EchoDoppler is the reference method for assessment of aortic stenosis and provides prognostic elements. However, it is imperfect with many inconsistencies between measures. On the other hand, the prognosis of patients with low flow and low gradient aortic retraction is discussed.

The main objective of this work is to study the prognosis of asymptomatic and symptomatic aortic retraction.

DETAILED DESCRIPTION:
Aortic stenosis is an attack most often acquired from the aortic valve corresponding to a defect of opening of this valve. Its prevalence increases with age and approaches 2% at age 65 and 25% at age 85 . It is in the majority of cases degenerative due to the development of calcifications on the aortic sigmoid valves by a process close to atherosclerosis (Otto CM, Circulation, 1994). It is associated with cardiovascular risk factors (age, male sex, smoking, high blood pressure and associated high LDL cholesterol). Aortic stenosis may also frequently be the consequence of aortic bicuspid (congenital) or more rarely rheumatic fever.

Aortic stenosis is responsible for an obstacle to ejection of the left ventricle with increased afterload and thus left ventricular work. After a long asymptomatic period when the obstacle to ejection is compensated by the induction of an adaptive left ventricular hypertrophy, symptoms appear initially of effort (dyspnea, angina, lipothymia see syncope) then clinical signs of insufficiency heart. The occurrence of symptoms should cause aortic valve replacement because at this stage the prognosis becomes unfavorable with a risk of death by cardiac decompensation or sudden death.

The two pillars of the diagnosis of severity are the evaluation of functional aortic valve area and the average transvalvular gradient. The tight aortic stenosis is defined for a functional aortic area <1cm² or 0.6cm² / m² and a mean tranvular gradient> 40 mmHg.

Patient survival data and / or a possible complication or indication for surgery will be evaluated periodically either during a standard follow-up consultation if patients are followed in the referral center or by telephone contact with the attending physician or cardiologist. . In case of death, the cause and date will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Retrospectively, all patients examined from January 1, 2000 to November 2014 will be included in the echocardiography laboratory whose objective examination is a narrowing of the aortic valve (maximum transaortic velocity ≥2.5 m / s).
* Aortic stenosis may be known in the past.

Exclusion Criteria:

* Refusal of the patient to participate in the study.
* Patients who have previously had aortic valve surgery before being examined in the echocardiography laboratory.
* Patients who can not be contacted or who do not respond will not be included in the database.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be identified from the transthoracic echocardiography reports of the echocardiography laboratory of CHU Amiens and CH Saint Philibert for the retrospective part. They are prospectively identified during echocardiography performed in the echocardiography laboratory of the two participating centers when a diagnosis of aortic stenosis is made. Patients will be informed by newsletter.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Prognosis of asymptomatic and symptomatic aortic valve stenosis | 6 years
  Aortic valve stenosis (Rao) is the most common valvulopathy in Western countries. Cardiac EchoDoppler represents the reference method of evaluation of Rao and provides prognostic elements. However, it is imperfect with many inconsistencies between measures. On the other hand, the prognosis of patients with low-gradient and low-gradient Rao is discussed.) The main objective of this work is to study the prognosis of asymptomatic and symptomatic aortic valve stenosis. To Look for predictors of prognosis and To Evaluate the impact of comorbidities on the prognosis of RAo Evaluate operative indications and specify the short and long term outcome after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe TRIBOUILLOY, MD, PhD, Principal Investigator — CHU AMIENS
Locations (1):
- Chu Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No